CLINICAL TRIAL: NCT06752200
Title: AMOUNT OF INTRAORAL OCCLUSAL ADJUSTMENTS IN OCCLUSAL SPLINTS FABRICATED USING FULLY DIGITAL VERSUS COMBINED DIGITAL WORKFLOW IN TMD PATIENTS (RANDOMIZED CONTROLLED TRIAL)
Brief Title: AMOUNT OF INTRAORAL OCCLUSAL ADJUSTMENTS IN OCCLUSAL SPLINTS FABRICATED USING FULLY DIGITAL VERSUS COMBINED DIGITAL WORKFLOW IN TMD PATIENTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma abd el fattah abbass sayed tantawy, Teacher assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D Ro 3_3_1
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: TMD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal splints fabricated using a fully digital workflow including the use of a jaw tracking devic (Experimental): The intervention involves the fabrication of 3D printing of occlusal splint with fully digitalization technique by the aid of Jaw Tracing Device (Zebis JMA, Germany).
  Interventions: Device: Occlusal splints fabricated using a fully digital workflow including the use of a jaw tracking device.
- Occlusal splints fabricated using a combined digital workflow using a conventional bite technique. (Active Comparator): For the comparator group, upper and lower arches will be scanned intraorally. The bite will be registered at centric by using rubber base bite registration material after patient deprogramming with Lucia jig. Then the bite will be scanned. The splint will be designed and printed in the same workflow as the intervention group.
  Interventions: Device: Occlusal splints fabricated using a combined digital workflow using a conventional bite technique

INTERVENTIONS:
Device: Occlusal splints fabricated using a fully digital workflow including the use of a jaw tracking device. — Occlusal splints fabricated using a fully digital workflow including the use of a jaw tracking device.
  Arms: Occlusal splints fabricated using a fully digital workflow including the use of a jaw tracking devic
Device: Occlusal splints fabricated using a combined digital workflow using a conventional bite technique — upper and lower arches will be scanned intraorally. The bite will be registered at centric by using rubber base bite registration material after patient deprogramming with Lucia jig. Then the bite will be scanned. The splint will be designed and printed in the same workflow as the intervention group.
  Arms: Occlusal splints fabricated using a combined digital workflow using a conventional bite technique.

SUMMARY:
Each eligible patient will be randomly into one of two groups:

group A: Occlusal splints fabricated using a fully digital workflow including the use of a jaw tracking device.

group B: Occlusal splints fabricated using a combined digital workflow using a conventional bite technique.

The intervention involves the fabrication of 3D printing of occlusal splint with fully digitalization technique by the aid of Jaw Tracing Device (Zebis JMA, Germany). The acquisition and scanning of the patients are done by using an intra oral scanner (Medit i700, South Korea) and designing them using a designing software (Exocad, USA). This device will be printed with a 3D printer (Anycubic, China) utilizing printable resin material with codes for which the outcome assessor is kept totally unaware.

For the comparator group, upper and lower arches will be scanned intraorally. The bite will be registered at centric by using rubber base bite registration material after patient deprogramming with Lucia jig. Then the bite will be scanned.

The splint will be designed and printed in the same workflow as the intervention group.

The amount of intraoral occlusal adjustments (represented by the 3-dimension volumetric changes) will be measured by Medit link by millimeters before the splint insertion.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18-40 years old

  (2) Complete dentition.

  (3) Normal jaw opening.

  (4) Intact teeth.

  (5) No occlusal disorder; stable jaw relation.

  (6) No ongoing dental therapy, such as orthodontic or prosthodontic treatment.

  (7) TMD patients with more than one of following symptoms or signs: myofascial pain and /or pain in the TMJ, myofascial pain and/or pain in the TMJ on palpation, muscles tenderness, headache or earache.

  (8) Patients who had unsuccessfully undergone splint therapy or other TMD treatments in the past were not excluded.

Exclusion Criteria:

* (1) Patients with an unstable occlusion

  (2) Patients with systemic diseases and comorbidities

  (3) Temporomandibular joint lesions found on clinical palpation or medical imaging examination

  (4) Jaw opening less than 3 fingers

  (5) Patients with occlusal dysfunctions

  (6) Patients with severe or moderate periodontitis

  (7) Unable to undergo examination or treatment due to the presence of a psychological or mental disorder.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The amount of intraoral occlusal adjustments (represented by the 3-dimension volumetric changes) | 5 weeks

IPD SHARING:
Plan to Share IPD: No
I am not going to share the IPD for privacy and security of the informations